<u>Title:</u> Promoting Asthma Guidelines and Management Through Technology-Based Intervention and Care Coordination (PRAGMATIC)

NCT03066596 IRB#: 2016-6258

IRB Approval Date: 11/06/2020

## **CONFIDENTIALITY STATEMENT**

This document is confidential communication. Acceptance of this document constitutes agreement by the recipient that no unpublished information contained herein will be published or disclosed without prior approval of the Principal Investigator or other participating study leadership and as consistent with the NIH terms of award.



# Promoting Asthma Guidelines and Management through Technology-Based Intervention and **Care Coordination (PRAGMATIC)**

#### Investigators:

Marina Reznik, MD, MS - PI Jill S. Halterman, MD, MPH Michael Rinke, MD, PhD Suzette Oyeku, MD Deepa Rastogi, MBBS Bruce Rapkin, PhD Sande Okelo, MD, PhD Cheng-Shiun Leu, PhD

## **Background**

Asthma disproportionately affects low-income and minority children residing in inner cities such as the Bronx, NY.<sup>1,2</sup> Use of national guidelines reduces asthma morbidity by 70%<sup>3</sup>; yet, these guidelines are not consistently implemented.<sup>4-11</sup> For example, providers' failure to document symptom severity and control in the medical record can lead to inadequate prescription of controller medications.<sup>42</sup> Providers also often fail to assess patients' inhaler technique, 10 identify in-home exposures, 43 and evaluate asthma co-morbidities. 44-46 Asthma education and action plans are not consistently provided. 42, 47-49 System-level barriers found in our research include limited access to resources (e.g. sample MDI-spacers) necessary to follow the recommended care. 10 Provider-level barriers include lack of awareness, disagreement with the guideline recommendations, lack of self-efficacy for being able to carry out the best practice, low expectation that outcomes will improve, and external barriers such as time constraints during a visit. 6, 7, 10 Patient factors may affect adherence to preventive medications. Many parents have uncertainty about the effectiveness of medications, lack understanding about proper use of preventive medicines and administration devices, and have concerns about potential side effects. 37, 49, 50 Other factors, such as financial barriers and problems with access to care have also been reported.<sup>51, 52</sup> There are missed opportunities to improve asthma care within the context of the child's medical home, particularly during clinic visits that are not asthma-related.<sup>26, 42, 53</sup> A recent AHRQ review of interventions to improve provider adherence to national asthma guidelines concluded that systems-level interventions that address barriers and all the elements of the asthma care process (i.e., prescription of controller medication, environmental control practices, self-management education, documentation of severity and control) are needed.9 Although interventions to improve provider adherence to asthma guidelines have been described. 12-24 few studies address translation of guidelines into routine care. 25, 26

The proposed translational study builds on our experience evaluating a Multifaceted Prompting Intervention (MPI) in 12 urban clinics.<sup>27</sup> MPI uses guideline-based prompts at the time of an office visit to support providers' decision-making, increasing the likelihood that they will recommend corrective actions (i.e., preventive medication prescription) to improve asthma management. We found that MPI delivered at one visit led to improved preventive care and short-term clinical outcomes (defined as number of symptom-free days (SFDs)).<sup>28</sup> Although effective, this intervention must be modified in several ways to translate into practice.

Our earlier study found that one-time prompting did not improve long-term clinical outcomes, so support at multiple visits is warranted. Further, MPI was implemented by the research team to a sample of children with persistent asthma. Successful translation means that guideline-based care is delivered by providers and staff to all children with asthma, rather than just a research sample. The prompt was printed on paper, rather than delivered through the electronic health records (EHR), limiting wide-scale adoption. Further, the original study did not offer support for caregivers to follow through on providers' recommendations (e.g., filling prescriptions, ongoing self-management, medication adherence). Although providers are directly responsible for making healthcare recommendations to patients, delivery of guideline-based care requires all clinic staff to facilitate

communication, make changes to clinic work flow, and ensure patients and caregivers are able to follow recommended corrective actions. In order to translate MPI to pediatric practices, we will enhance it in several ways: (1) use clinic rather than research staff to facilitate assessment for prompts at every visit; (2) ensure prompting for guideline-based care for all children ages 2-12 with persistent or uncontrolled asthma, rather than just a research sample; (3) routinely deliver prompts to the provider via EHR; (4) offer telephone-based care coordination, education and support to children with the highest morbidity via a dedicated Outreach Worker (OW) to ensure recommendations are followed; and (5) provide practice-level supports (e.g. clinic champions, on-going performance feedback and participatory problem solving) to promote full adoption of guidelines. The enhanced MPI program (eMPI) consists of innovative multi-level and team-based strategies to enable providers to effectively and efficiently adopt asthma care guidelines.

We will conduct a cluster randomized trial comparing eMPI to enhanced usual care (eUC) in 22 Bronx practices serving over 5,000 children ages 2-12 years with persistent or uncontrolled asthma. Eleven eUC practices will receive guideline information and assess children's asthma severity and control, but active intervention components will not be provided. Practices will join the study in 4 waves over 4 years (4-6 practices per year). Including attendings and residents we anticipate enrolling an estimated 200 providers into the study.

# **Study Objectives**

This study has the following objectives:

- 1. To test the impact of eMPI on provider adoption of asthma management guidelines. The primary outcome is a clinic-level variable measured by the proportion of visits with >1 guideline-based corrective actions, as indicated in the EHR (i.e., controller medication prescription or adjustment, trigger evaluation). In this analysis we will include all patients ages 2-12 years with persistent or uncontrolled asthma (~5,000). Hypothesis 1 (primary): eMPI will improve provider adoption of asthma guidelines compared to eUC.
- 2. To determine whether consistent use of eMPI leads to both short- and long-term improvements in clinical outcomes. Our main clinical outcome is improvement in SFDs. Since these data are not in the EHR. we will randomly sample 512 children's caregivers from eMPI and eUC practices. Caregivers will be interviewed every 3 months to examine short- (at 3 months) and long-term (at 6-12 months) change in SFDs. Hypothesis 2a (secondary): Short- and long-term improvements in SFDs will be greater in eMPI over eUC. Hypothesis 2b (secondary): We also will assess if these improvements are mediated by corrective actions taken at the visit.
- 3. To evaluate the process of program implementation. We will apply the RE-AIM framework to address the intervention's Reach (the provider-level proportion of visits with corrective actions), Effectiveness (provider corrective actions and SFDs), Adoption (the pace and level of uptake of quidelines), Implementation (improvements in reach and effectiveness over successive waves), and Maintenance (sustainable use of guidelines). We will evaluate group differences in the extent of healthcare utilization and resources used (i.e., adherence to clinic follow-up visits, specialty referrals, emergency and in-patient care, OW referrals).

## Study Overview

#### A. Study Design

Design Overview: We will conduct a 2-group cluster randomized trial comparing eMPI to enhanced usual care (eUC) in 22 Bronx practices serving over 10,000 children with asthma. The randomization will be at the practice level to avoid contamination. Each practice will be matched into 11 similar pairs based on size and type and then randomly assigned to either eMPI or eUC.

Provider adoption of guidelines and utilization of care in all patients (~5,000) ages 2-12 years with persistent or uncontrolled asthma from eMPI and eUC practices will be evaluated using EHR data and practice-based screening for asthma severity and control. We will also enroll a random subset of 512

caregivers of children with persistent/uncontrolled asthma from both study arms to systematically evaluate caregiver-reported child morbidity outcomes and obtain measures not available in EHR. These children will be enrolled at the time of the office visit and followed prospectively for 4 time points - 3, 6, 9, and 12 months after the initial visit - to assess clinical and process-focused outcomes.

## **B. Subjects and Setting**

Outpatient practices (n=22) that are part of Montefiore Health System will participate in the study (see Letter of Support). These 22 practices are located throughout the Bronx, NY, represent different practice types, and have participated in several of our prior studies (Table 3). Though there were initially 22 proposed outpatient practices, two practices were closed, two practices (FCC-B and FCC-C) were combined as a single site given that they serve patients in the same facility, and one practice was excluded given no pairing available, resulting in a total n=18 participating outpatient practices. The number of children with asthma across practices (N=10,109) of whom we estimate ~ 50% (N=5,000) to have persistent or

| Table 1. Primary Care Practices* | | | | | |
|---|---|---|---|---|---|
| Site | Practice Type | Provider Type | # 2-12yr olds<br>in practice | # 2-12yr olds<br>with asthma | # visits for 2-<br>12yr olds with<br>asthma |
| Astor Avenue | NHC | Pediatrics | 3,075 | 576 | 1,012 |
| Bronx East | NHC | Pediatrics | 4,775 | 884 | 1,516 |
| Burke Avenue | NHC | Pediatrics/Family MD | 1,102 | 117 | 196 |
| Castle Hill | FQHC | Family MD | 814 | 97 | 135 |
| CFCC | FQHC | Pediatrics | 5,791 | 1,144 | 1,824 |
| CHCC | FQHC | Pediatrics | 4,658 | 1,332 | 2,488 |
| Co-op Bartow Ave | NHC | Pediatrics | 2,485 | 634 | 1,059 |
| Eastchester | NHC | Pediatrics | 1,350 | 325 | 703 |
| FCC - B | Hospital Clinic | Pediatrics | 3,671 | 684 | 1,028 |
| FCC - C | Hospital Clinic | Pediatrics | 3,470 | 805 | 1,300 |
| FHC | FQHC | Family MD | 1,739 | 339 | 606 |
| Grand Concourse | NHC | Pediatrics/Family MD | 3,133 | 540 | 868 |
| Grand UCC | NHC | Pediatrics/Family MD | 2,950 | 235 | 262 |
| HIP Cross County | NHC | Pediatrics/Family MD | 3,058 | 272 | 385 |
| MAP-8 | Hospital Clinic | Pediatrics | 2,935 | 631 | 1,551 |
| Marble Hill | NHC | Pediatrics/Family MD | 1,143 | 186 | 294 |
| University Avenue | FQHC | Pediatrics/Family MD | 1,697 | 344 | 645 |
| Verde Clinic | NHC | Family MD | 359 | 78 | 146 |
| Wakefield | NHC | Pediatrics | 354 | 309 | 600 |
| West Farms | FQHC | Family MD | 954 | 215 | 368 |
| White Plains Road | NHC | Pediatrics/Family MD | 1,204 | 174 | 273 |
| Williamsbridge | FQHC | Family MD | 1,059 | 188 | 308 |
| TOTAL | - | - | 51,776 | 10,109 | 17,567 |

T QTIO-1 edetaily Qualified Treatile Center, 14 TO-14 egistori food feature Center. Trainible of patients 3 eem between 17 1714-123 1714

uncontrolled asthma is sufficient to meet our sample size needs. A subset of 512 children will be recuited over 4 years (~128 participants each year) to obtain clinical outcomes data that are not in the EHR.

**Randomization:** Prior to participant enrollment, each practice will be matched into 11 pairs based on size of the practice and provider type (Table 1). Practices will then be randomly selected within each pair as an eMPI or a eUC site. Practices will join in 4 waves over the course of 4 years (4-6 practices/year). Each practice will remain in the study for 24 months and receive \$500 donation to thank them for participation.

*Inclusion Criteria:* The criteria listed below will apply to ~5,000 children from eMPI and eUC practices. We will obtain a waiver of consent to be able to review EHR data by practice.

- (1) Physician-diagnosed asthma (based on EHR).
- (2) Persistent or uncontrolled asthma as per clinic assessment. Based on NHLBI guidelines,  $^{41}$  any one of the following: in past month, > 2 days/week with asthma symptoms, > 2 days/week with rescue medication use, > 2 days/month with nighttime symptoms, or > 2 episodes in the past year that required systemic corticosteroids.
- 1) Mild persistent or more severe asthma severity, or poor asthma control (see definitions below). \*A different assessment of eligibility will be performed depending on whether or not the child has a current prescription for preventive asthma medication at baseline and parent reports its use. This is consistent with the EPR recommendations that make a strong distinction between classifying asthma severity (for children not using preventive medications) and assessing control (for children using preventive medications). If a child has used a preventive medication in the past, but reports no use of the medication in the prior 3 months, we will assess severity. This 3-month time frame is consistent with the length of "wash-out" time for inhaled steroids. 152
  - a) **Children not using a preventive medication at baseline**: Mild persistent to severe persistent asthma.<sup>9,10</sup> Any 1 of the following, during the prior 4 weeks (as defined by parent interview in the waiting room and EMR review):
    - i) An average of >2 days per week with asthma symptoms
    - ii) >2 days per week with rescue medication use
    - iii) ≥3 nights per month awakened with nighttime symptoms
    - iv) Minor limitation of activity
    - v) >2 episodes of asthma during the past year that have required systemic corticosteroids
  - b) **Children using a preventive medication at baseline**: Poor asthma control. Any 1 of the following, during the prior 4 weeks (as defined by parent interview in the waiting room):



- i) An average of >2 days per week with asthma symptoms
- ii) >2 days per week with rescue medication use
- iii) >2 nights per month awakened with nighttime symptoms
- iv) Some limitation of activity
- v) >2 episodes of asthma during the past year that have required systemic corticosteroids.
- (3) Age 2 and 12 years, inclusive.

Additional inclusion criteria will apply to a subset of 512 of children whose caregivers will be interviewed to systematically evaluate experiences with the program and caregiver-reported morbidity outcomes:

- (1) Caregiver is able to speak and understand either English or Spanish. Participants unable to read will be eligible as all surveys will be administered verbally by research personnel.
- (2) Consent from the primary caregiver, caregiver permission for the child to participate as well as assent from the child (>7 years). If there are eligible siblings, they will be enrolled if logistically possible.

## Exclusion Criteria:

(1) The child has other significant medical conditions, such as congenital heart disease, cystic fibrosis, or other chronic lung disease, that could interfere with the assessment of asthma-related measures.

Additional exclusion criteria will apply to a subset of 512 children/caregivers as described above:

- (1) No access to a telephone to conduct follow-up surveys.
- (2) Children in foster care or other situations in which consent cannot be obtained from a quardian. Based on our previous studies, we anticipate <10% of children will be excluded based on these criteria.

Screening: In 22 practices, clinic staff (RN/LPN) will ask caregivers of all children 2-12 years of age with asthma to complete a screening survey in EPIC Electronic Health Record (EHR) during the triage portion of their doctor visit. The screening survey questions follow national guidelines and will identify children with persistent or uncontrolled asthma (Appendix A).

Procedures for enrollment of a subset (n=512): Clinic staff will inform research team on days of recruitment to obtain consent and baseline assessment from a subset of children with persistent or uncontrolled asthma and their caregivers from whom additional morbidity measures (not present in the EHR) will be collected. Enrollment goals for each practice will be based on the number of children with asthma seen at the practice. Since enrollment will occur over an extended time period, we will block enrollment by site pair to assure an equal balance of children in each group for each seasonal time period. Research staff will be present in each clinic 2-3 days/week for recruitment, until monthly enrollment goals are met for that practice. We will review the practice's schedule the day before to determine if potentially eligible participants are scheduled for a visit. Research staff will call patients with asthma ages 2-12 years and ask families to come to their appointment with physician 30-60 minutes earlier to be screened by the nursing staff for asthma severity. If eligible, the caregiver/child will be informed about the study, undergo the informed consent process and complete baseline survey prior to seeing the physician. Recruitment goals will be reviewed weekly for each practice and adjustments of staffing made as needed. Days for recruitment will vary to ensure that patients of providers who are in clinic on certain days of the week are not over- or under-sampled (see Recruitment Protocol, Appendix A). Following informed consent/assent, research staff will conduct a 10-minute survey with the primary caregiver in the waiting room to obtain baseline measures of enrolled participants. All survey instruments will be available in English/Spanish and questions will be read aloud. Caregivers will be offered a private location within the waiting room to complete the survey. The baseline measures include standard demographic and health history variables, healthcare utilization, quality of life, beliefs about medication and adherence (Appendix A).

IRB NUMBER: 2016-6258 IRB APPROVAL DATE: 11/06/2020

**eMPI Intervention:** The eMPI components are described in Table 4 and closely mirror implementation strategies recommended by the panel of experts in implementation science for development of a tailored multilevel strategy for implementation.<sup>54</sup> First, at every office visit, caregivers of children ages 2-12 years with persistent or uncontrolled asthma will be asked to complete a screening survey in EPIC Electronic Health Record (EHR) during the triage portion of their doctor visit (Appendix A). Clinic staff will review the answers with the caregiver and read the questions aloud as needed. Based on these responses, a prompt for both the provider and caregiver will be generated in EPIC EHR using a simple algorithm (Appendix B). The provider prompt will be delivered to the provider at each visit via EHR and include information on child's current level of asthma severity or control, controller

#### TABLE 4. CORE ELEMENTS OF eMPI MULTI-LEVEL TRANSLATIONAL STRATEGIES

#### Direct Support for Providers' Delivery of Guideline-Based Care in Practice

- Caregiver waiting room assessment of asthma severity and control
- Provider prompts to deliver guideline-based corrective actions at every visit
- Caregiver prompts to encourage discussion with provider
- Enhancements to Increase the Feasibility and Sustainability of eMP
  - Waiting room assessment for the prompts on Tablet PCs
  - Physician prompts in Electronic Health Record (EHR)

#### Involving Clinic Staff in Promoting and Supporting Use of Guidelines

- Regular staff administer and survey information for prompts
- Outreach Worker-delivered care coordination and support to ensure recommendations are followed by patients

#### Building Accountability and Commitment to Guideline-Based Care

- Designation of clinic champion to lead practice change
- Designation of Practice Advisory Board to monitor and guide change

### Promoting Providers' Understanding, Acceptance and Use of Guidelines

- Interactive seminars about asthma guidelines, pocket cards with guidelines
- Ongoing feedback about performance improvement
- Identification of barriers to guideline use and eMPI implementation
- Ongoing sharing of best ideas and solutions to overcome barriers

medication use, exposure to triggers, and specific tailored recommendations for guideline-based preventive care (e.g. for persistent asthma without controller medication, the recommendation on the prompt will include starting controller medication).<sup>41</sup> For children with poor control despite being on controller medications, recommendation will include evaluation of inhaler technique and medication adherence, treatment and referral for evaluation of co-morbidities (e.g., referral to the Asthma Center for allergy and pulmonology consultations), "step-up" of medications, evaluation and counseling on triggers, and outreach worker referral (See below). The prompt will also include a recommendation for the provider to establish treatment goals with the patient and inquire about any caregiver's concerns. The prompt for the provider will be seen on the computer screen in EPIC EHR at the time of the visit allowing provider to check off the guideline-based recommended items discussed during the visit. The caregiver prompt will include immediate feedback on child's asthma severity/control with personally tailored information highlighting caregiver's goals and concerns. The prompt will include simplified recommendations for preventive care issues to discuss with the provider during the visit (e.g., to discuss triggers, medication concerns, need for asthma action plan (AAP) and medication administration form (MAF) for school). AAP and MAF are embedded into EPIC EHR patient chart and can be printed and given to patient to take home or to school. The caregiver prompt is based on the guideline recommendation to promote joint discussions about treatment plan and goals and will be printed for caregiver to bring to the visit. Outreach worker (OW)-delivered telephone-based care coordination and support will be provided by the bilingual (English/Spanish) OWs, lay people from the community who have asthma or a child with well-controlled asthma. OWs will become a practice-based resource. OWs will provide telephone-based care coordination, education and support to children who are already on controller medication but still have uncontrolled asthma and other barriers to guideline-based care (e.g., unable to fill a prescription, loss of medical insurance, poor medication adherence, gaps in caregiver knowledge despite provider education). The decision to refer family to OW service will be based on provider's assessment at any office visit. Providers will be prompted to make OW referrals for children with uncontrolled asthma as part of the guideline-based care. We estimate that 20% of children in each intervention practice will be referred to the OW. Providers will have a referral mechanism embedded within EHR to refer patients to the OW with suggestions on which children should be referred. OW training: OWs will be trained (4-weeks) by the PI (Reznik) and Co-Is (Rastogi, Jariwala) using evidence-based guidelines on asthma self-management skills, proper inhaler technique, triggers, medication use, goal setting and problem solving. The PI will oversee OWs with bi-weekly (and more often if needed) meetings to discuss cases/concerns and will listen to 20% of the recorded telephone calls to ensure the OWs deliver the sessions as intended. OWs role: OWs will help facilitate implementation of the guideline-based care prescribed by provider at the office visit. If referred to the OW at the initial visit, the first OW telephone call with the child's caregiver will occur within 2 weeks after the initial visit to determine any care coordination needs (e.g., assistance scheduling specialty appointments, inability to fill prescriptions) and then monthly, starting at 1-month post-initial visit for 6 months. If referred at the follow-up office visit, the same

IRB NUMBER: 2016-6258
IRB APPROVAL DATE: 11/06/2020

schedule of OW calls will apply. OWs will use evidence-based educational materials that were previously adapted to the needs of our community, and focus on helping parents develop 6 key asthma management behaviors as per NHLBI guidelines<sup>41</sup> and our prior research using OWs: (1) Asthma control monitoring, (2) Identifying and minimizing exposure to triggers, (3) Effectively using controller medications, (4) Using quickrelief medications, (5) Using an asthma action plan, and (6) Effectively working with the child's physician and schools on optimizing asthma care. The decision to work on specific behaviors will be tailored to caregiver needs expressed at the provider visit and based on caregiver's concerns and goals identified by the caregiver prompt. During the telephone calls. OWs will also assist with patient care activities (e.g., scheduling appointments, refer to community services for Integrated Pest Management provided by the NYC Department of Health, smoking cessation programs (NYS Smokers' Quitline), free legal services and existing on-line resources) and share information with the provider and other members of the clinical team via EHR if any concerns about patient or caregiver arise during the telephone encounters (e.g., caregiver does not have prescription for medication, child seen in ED or hospitalized). The OWs will use a Microsoft Access database to record call frequency, length, and notes taken. These calls will last ~30 minutes. OWs will also send text messages, if preferred by the caregivers, to remind about clinic appointments or schedule follow-up telephone calls.

**Translational Process within eMPI Clinics:** At each intervention clinic, there will be three phases of eMPI translation into routine practice: 1) *initiation* (3 months, intense support provided), 2) *consolidation* (3 months,



support available), and 3) *sustainability* (18 months, support as needed). During the *initiation* phase, the goal will be to introduce eMPI to the practice. First, we will partner with a *clinic champion*, a practice physician who

will also serve on our *Practice Advisory Board*. The Board will consist of > 2 physicians, 1-2 nurses, 1-2 front desk and administrative staff. The Board will meet monthly during the initiation and consolidation phases to review the study protocol as it relates to the practices, discuss any provider-reported barriers to implementation and identify solutions to address these barriers using a collaborative problem solving approach. These Boards will capitalize on already existing and engaged groups created by the Bronx Ongoing Pediatric Screening in the Medical Home (BOPS) program described in the Preliminary Studies section. To initiate the planning process, we will ask Board members to complete the RE-AIM planning tool96 to highlight any concerns or barriers to implementation. We will engage providers in a practice improvement process by having the clinic champion discuss feedback received from individual providers and solutions at the regular clinic meetings. We will provide the champion with a tool, updated monthly, to record identified barriers to guideline implementation and ways to address them. We will also collect baseline information on provider corrective actions in EHR; assess provider self-efficacy, provider-caregiver communication, and provider competencies in guidelinebased care using a validated survey (Appendix A). During month 1 of the initiation phase, we will provide practice-level support (e.g., pocket cards with quidelines, brief interactive seminars, local asthma resources; Appendix C) to the practices to assist providers in implementing the asthma management outlined in the NHLBI guidelines<sup>41</sup> and to help remove practice and provider-level barriers to guideline implementation.<sup>7, 10</sup> The interactive seminars, developed using principles of physician behavior change<sup>97</sup> and led by the PI (Reznik) and co-ls (Rastogi, pulmonologist and Jariwala, allergist), will generate enthusiasm around prompting and empower providers to implement desired changes. The seminars will include an overview of guideline-based asthma care and orientation to the prompts, resource guides and the feedback charts. At the end of the seminar, a brief needs assessment survey will be done, and additional resources will be provided based on the needs of the individual practices. Providers will receive continuing education credit for their participation. These sessions will be coordinated by each practice's champion. We will also provide practice-level feedback. eMPI practices will receive monthly feedback during the initiation phase on the proportion of visits with appropriate guideline-based preventive actions, and the proportion of patients meeting goals of therapy (limited symptoms, no ED visits/hospitalizations). The feedback will be delivered to the champion who will then share it with the rest of the providers. The information will be presented graphically with other intervention practices displayed by a code for comparison. A Quality Control Tool will be used to measure and assess nurse adoption of the asthma severity/control screening. Research staff will observe nursing staff at least once during the

6

EINSTEIN IRB NUMBER: 2016-6258

implementation period as they conduct the severity/control asthma screening, make note of their screening practices and provide feedback to the nursing staff and the clinic champion. During the consolidation phase, we will continue to work with site champions and practices to ensure eMPI is implemented as intended and provide support on addressing barriers or concerns. Major activities during this time will include on-going monitoring of all aspects of eMPI, feedback to sites about their performance, identification of barriers and needed resources, and Board meetings to address these impediments. Given the COVID-19 pandemic, as of March 2020, Board meetings have been restricted to telephonic or video conference call only. We will finalize a sustainability plan with each practice to ensure on-going use of guidelines. During sustainability phase, we will observe practices' continued use of guideline-based care. During this time, we will not provide regular consultations or support, but will be available to address questions and concerns that arise. This will allow us to monitor how much outside help sites require to sustain eMPI. We will provide feedback at the practices' request. We expect that eMPI practices undergoing our translational program will increase guideline-based care during a 3-month initiation period and subsequent 3-month consolidation period, and will maintain these gains over an 18-month sustainability period.

Enhanced Usual Care (eUC) Practices will receive a review packet of the NAEPP quidelines<sup>41</sup> and educational resources for families. Children will be assessed for asthma severity and level of control at each visit as best-practice care, but active intervention components will not be provided.

Outcomes Assessment. Follow-up assessments for 512 participants will be conducted by interviewers blinded to the treatment allocation at 3, 6, 9, and 12 months. Outcome measures will be assessed by telephone interview, and EHR data will be reviewed for all patients with asthma in both study arms. Given the minimal risk of survey questions and the importance of having full datasets for study analyses, in the case that study personnel are unable to reach the caregiver who signed consent at enrollment (after multiple phone attempts, letters, home visits, and scheduled appointment outreach), we will proceed to obtain verbal consent and survey data from another caregiver who is aware of the enrolled child's history with asthma. These caregivers include the other parent, guardian, grandparent, aunt, or uncle. Name and contact information of the alternate caregiver will have been provided at enrollment by the caregiver who initially signed consent.

**Measures:** The following measures are organized by clinic-, provider- and patient-level variables.

### Clinic-Level Variables

The *primary outcome* is a clinic-level variable measured by the proportion of visits with >1 guideline-based corrective actions. To calculate this proportion, the denominator will include only the visits by patients aged 2-12 years with persistent or uncontrolled asthma at the time of visit. We will obtain these data from the EHR at baseline, monthly during the initiation phase (to provide feedback to eMPI practices) and every 3 months thereafter for 24 months. Corrective actions include: (1) prescription of a new preventive asthma medication; (2) increase in dose of a preventive medication (for children already on preventive medication); (3) evaluation and counseling regarding triggers; (4) treatment of co-morbid conditions (e.g., sinusitis, allergic rhinitis, obesity); (5) referral to an allergy or pulmonary specialist. We will consider children receiving any of these guideline-based preventive care measures during the visit as having a corrective action (as not all actions may be necessary for each patient), and also will consider each component of preventive care separately. We collected prospective data on most items included in the corrective action definition in our prior work.<sup>28, 98</sup> Additional corrective actions include recommendations for a follow-up visit specifically to discuss asthma. referrals made to OW, and provision of an asthma action plan or school medication administration form. Covariate: Practice characteristics will include practice size (small, medium, large), practice type (hospitalbased practice, Federally Qualified Health Center, neighborhood health center), and patient mix (pediatrics, adult/pediatrics), involvement of support staff in the delivery of preventive asthma care, practice-level changes (e.g., new asthma-related initiatives in the practice). We will obtain this information from the existing database of practices and from interviews with the physician champion and office administrator at each practice.

### **Provider-Level Variables**

Potential Mediators: 1) Provider Competencies: We will assess a) provider's asthma practices (frequency of assessing patient symptom severity, treatment adherence, and use of guideline-consistent care), 99, 100 and b)

frequency of use of communication and education strategies contained in the Physician Asthma Care Education (PACE) physician survey. 101 2) Provider/Caregiver Communication: We will ask providers in all practices to complete a brief survey at the beginning (during initiation) and end of the study (during sustainability phase). The survey is adapted from the PACE<sup>102</sup> assessment and includes questions about asthma care practices and communication with families. The providers will also be asked if they have been involved in other quality improvement or educational efforts on asthma care. Survey link will be sent to providers electronically.

Covariate: We will collect data on provider type (MD. PNP, PA), the level of training (resident or attending). specialty (family medicine or pediatrics), and if the visit's provider was the child's primary care provider. We will obtain this information from the chart review, caregiver interview for a subset of patients and provider survey.

#### Patient-Level Variables

Clinical/Functional Outcomes will be collected from caregivers of 512 children (Table 5).

1. Asthma Symptoms: We will assess number of symptom-free days (SFDs) (secondary outcome measure) at baseline. 3 months to determine shortterm effectiveness of the intervention. and at 6, 9, and 12 month follow-up evaluations to assess long-term intervention effects. This outcome

| Table 5. Measures | Measurement Strategy | Time of Administration |
|---|---|---|
| Clinical/Functional Outcomes | | |
| Asthma Symptoms | Caregiver report on SFDs, ACT, <sup>105</sup><br>NHLBI guidelines <sup>41</sup> | Baseline; 3, 6, 9, & 12 months |
| Healthcare Utilization | Caregiver interview on health care contacts; EHR data | Baseline; 3, 6, 9, & 12<br>months; chart review |
| Quality of Life | Caregiver interview – Juniper Scale <sup>106</sup> | Baseline; 3, 6, 9, & 12 months |
| Functional Severity | Caregiver interview – Child Health<br>Survey for Asthma <sup>107</sup> | Baseline; 3, 6, 9, & 12 months |
| Medication Beliefs/Adherence | Caregiver interview – Horne Scale <sup>108</sup> | Baseline; 3, 6, 9, & 12 months |
| SFDs=Symptom-Free Days; ACT=Asth | ma Control Test; EHR=Electronic Health Records | |

measure is consistent with the symptom monitoring recommended by the national guidelines and has been suggested as a useful endpoint for pediatric asthma studies. 103, 104 Caregivers will be asked to report the number of days their child experiences no symptoms of asthma (defined as 24 hours with no coughing, wheezing, chest tightness, or shortness of breath) in the past 2 weeks. We will also assess asthma control with the Asthma Control Test. 105

- 2. Healthcare Utilization: Caregivers will report child's healthcare utilization at baseline and each follow-up. In addition, EHR data will be reviewed at each follow-up to assess for office visits (acute and routine), emergency department visits and hospitalizations. We will also evaluate healthcare utilization outcomes from the EHR data review for all patients with persistent or uncontrolled asthma (~5,000) across practices.
- 3. Quality of Life: Quality of life will be measured at baseline and each follow-up using Juniper's Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ). 106 The PACQLQ is a standard instrument used to assess the quality of life of caretakers of children with asthma, and provides a quantitative score that reflects answers to questions about the burden of caring for a child with asthma. 106
- 4. Functional Severity: Functional limitations of the child will be assessed at baseline and each follow-up evaluation using a subscale from the Children's Health Survey for Asthma. 107 The child activity subscale includes 5 items on limitations to the child's activities due to asthma (Cronbach's alpha .87-.89).
- 5. Beliefs about Medications and Adherence: We will use the 10-item Horne's Beliefs about Medications Questionnaire (BMQ).<sup>108</sup> Five questions assess parent's views about the necessity (alpha=.80) and five measure parental concern about their child's medications (alpha=.75). The 4-item Adherence Scale<sup>108</sup> measures parent-reported medication adherence using a 5-point Likert scale (alpha=.60-.83).

#### Covariates:

- 1. Demographic Variables will include child's age, gender, race, ethnicity, medical insurance, and caregiver's education level. We will use standardized questions from the national child health surveys to obtain these data.
- 2. Medical Variables will include birth history (prematurity), duration of asthma diagnosis and history of allergies (e.g., allergic rhinitis, seasonal allergies) or eczema.
- 3. Caregiver Depression: Caregiver depression has been shown to affect adherence to care plans, communication and child's asthma outcomes. 109, 110 We will assess maternal depression using a validated Patient Health Questionnaire 9 (PHQ-9).111

**EINSTEIN** IRB NUMBER: 2016-6258 IRB APPROVAL DATE: 11/06/2020

#### Potential Mediators:

- 1. Caregiver/Provider Communication: We will use 5 communication items from the PACE Parent/Caregiver Questionnaire<sup>102, 112</sup> to assess caregiver's perception of their communication with the provider. Items are scored on a 6-point Likert scale (Don't know, Strongly Agree-Strongly Disagree).
- 2. Self-Efficacy: We will assess caregiver self-efficacy in communication with their child's provider using the validated Perceived Efficacy in Patient-Physician Interaction questionnaire (PEPPI). 113-115

RE-AIM Measures: We will use RE-AIM framework<sup>93</sup> to evaluate the translational process: (1) the providerlevel proportion of visits with corrective actions (Reach); (2) the impact of the intervention on provider delivery of guideline-based care (corrective actions taken at the visit) and SFDs (Effectiveness); (3) the pace and level of uptake of guidelines and changes in service utilization (Adoption); (4) improvements in reach and effectiveness over successive waves (Implementation); and (5) continued use of guidelines and sustainability of strategies by practices in order to facilitate dissemination to other clinical settings (Maintenance). We will be completing post-study qualitative interviews with approximately 125 clinic stakeholders (e.g. advisory board members, physicians, medical directors, nurses, and administrative personnel) from both eMPI and eUC practices to further evaluate the process of program implementation. Individual interviews will be completed through Zoom audio conference call, where clinic stakeholders will answer questions related to their clinic's culture, asthma management workflows, and barriers and facilitators to program implementation. The interviews will be audio-recorded and transcribed verbatim for further qualitative analyses.

Analysis of qualitative data: Transcribed interviews will be imported into the NVivo qualitative data software to assist with data organization. Qualitative data will be analyzed according to the concepts of grounded theory. Codebooks will be developed in an iterative fashion. Coders will independently code the first 3 transcripts, meet to compare codes, and then alter or add codes as necessary. After this, a codebook will be created to include definitions, rules, and examples for each code. The coders will then code all subsequent transcripts and revise the codebook as necessary to incorporate new codes or refine existing codes. The constant comparison method will be used to determine if there are any patterns or themes by provider/stakeholder characteristics.

#### **Summary of Analytic Plan:**

We will use graphical and numerical summaries to describe the outcomes at each assessment point. If distributional assumptions for particular statistical procedures are violated, appropriate transformations will be made or non-parametric tests will be used. All primary and secondary analyses will follow the intent-to-treat principle; all participants will be analyzed in the group to which their clinic was assigned irrespective of their post-randomization behavior, and all participants will be analyzed using multiple imputation techniques. Hypothesis-driven comparisons will be made with control of the type I error rate at 0.05 (two-sided). Preliminary Analysis. We will examine data for out of range values. Descriptive statistics will be generated regarding practice characteristics such as size (small, medium, large), practice type (hospital-based practice, Federally Qualified Health Center, neighborhood health center), and patient mix (pediatrics, adult/pediatrics) to help to understand the sample as well as the generalizability of study findings. We will determine whether there are differences at baseline between the eMPI and eUC providers and patients in demographics and background characteristics. This will include analogs of t-tests (or Wilcoxon rank sum tests) for continuous variables and chi-square (or Fisher's Exact) tests for categorical variables adjusted by generalized estimating equation (GEE) methods for the clustering induced by providers within clinics.

## Aim 1. To test the impact of eMPI on provider adoption of asthma management guidelines.

The **primary outcome** is a clinic-level variable measured by the ratio of number of visits with >1 guidelinebased corrective actions to the number of visits by patients aged 2-12 years with persistent or uncontrolled asthma at the time of visit. The primary null hypothesis is that there is no difference between eMPI and eUC clinics in the mean proportion of visits where the necessary corrective actions were taken. To test this null hypothesis, we will use a matched-pairs randomization (or permutation test) at the 0.05 two-tailed level of

**EINSTEIN** IRB NUMBER: 2016-6258

significance. The permutation test will account for the fact that clinics (rather than providers) are randomized and that the randomization will be performed within clinic pairs. Each pair of clinics will produce a matched difference in the proportions of corrective actions, and under  $H_0$  the randomization can be viewed as attaching a random plus or minus sign. Thus there will be  $2^{11} = 2,048$  possible signed permutations, allowing a two-tailed p-value as significant as 2/2,048 < 0.001 (if all 11 pairs show a greater proportion of corrective actions taken by the eMPI practices). Assuming no important practice characteristics are significantly out of balance (at twotailed p<0.01), the permutation test will comprise the primary analysis. If any important clinic characteristics are significantly imbalanced at p<0.01, we will adjust for such variables in a linear regression model and report the adjusted intervention coefficient as the primary result. We will also examine for a clinic-size (or provider-type) by intervention interaction. If not significant at the 5% level, the above approach will be used to provide the primary results. If significant, we will attempt to identify factors that affect the primary outcomes and might differ between clinics (or provider types). If including such factors removes the interaction, we will quote the adjusted intervention effect from the model including such factors. If not, we will quote two intervention effects (for large and small clinics) leaving the interaction unresolved.

Power Analysis. We conservatively estimate that the mean difference between eMPI and eUC clinics in the proportion of visits where the necessary corrective actions were taken will be at least 25 percentage points. To express this as a standardized effect size, we assume the standard deviation of the paired differences in the proportion of corrective actions will be no more than 0.2, based on several mock data sets generated by the investigators reflecting their clinical experience and best estimates. We present one generated data set in Table 6 for illustration. This hypothetical data set has an average matched difference in proportions of 0.246 (about 25 percentage points) with standard deviation 0.142 (14.2 percentage points). Our assumption of a standard deviation of 0.2 or 20 percentage points is thus about 50% larger than in this illustrative example.

Table 6. A Mock Data Set

| Clinic Pair | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Proportion Difference | .25 | .10 | .20 | .50 | .00 | .25 | .30 | .40 | .10 | .30 | .30 |

The standardized effect size is therefore 0.25/0.20 = 1.25. Approximating the power of the permutation test by that of a paired t-test with 10 degrees of freedom, a sample size of 11 clinics per arm will yield a non-centrality parameter of 1.25√11 = 4.15, providing more than 95% power to detect a standardized effect size of 1.25 or more. The detectable effect size at 80% power is a mean difference 17.8 percentage points between eMPI and eUC practices. Even if the true standard deviation of the matched differences in proportions were as large as 0.281, we would still have 80% power to detect a 25 percentage point mean difference.

Aim 2. To determine whether consistent use of eMPI leads to both short- and long-term improvements in clinical outcomes. In this Aim, we will compare the change from baseline to each of the follow up (FU) time points (i.e., 3, 6, 9, and 12 months) in number of SFDs between eMPI and eUC patients using intent-to-treat principles. We will employ the generalized linear model (GLM) with identity link function for this comparison. The analysis model is of the form  $EY_{ij} = \alpha + \beta I_i + \sum \gamma_i T_{ij} + \sum \delta_i I_i T_{ij}$ , where for subject i  $Y_{ij}$  is the number of SFDs for at time j, li denotes group indicator for eMPI group (vs. eUC), and Tii is the indicator for time at FUj evaluation (vs. baseline). The regression coefficient  $\delta_i$  corresponding to the group-by-time interaction term estimates the difference in average change of SFDs at FUj evaluation vs. baseline, comparing eMPI to eUC groups, and thus represents the effect of intervention on the SFDs. We will use generalized estimating equations (GEE) methodology to account for within-subject correlation due to multiple assessments for the same subject as well as the within-provider and within-practice correlations due to cluster sampling. We will also determine whether or not the corrective actions taken mediates the effect of intervention on outcomes; we will use the test of joint significance of the 2 paths involving a potential mediator, which best balance Type I error and statistical power. 116 A variable M will be declared a mediator only if both the test of the regression coefficient of the explanatory factor X on the mediator and the test of the coefficient of the mediator on the outcome variable Y controlling for X are significant at level alpha = 0.05, 2-tailed. This approach allows for partial mediation which we fully expect to occur. In subsequent analyses we will estimate the indirect path effect with 95% confidence intervals using the asymmetric distribution of products method. 116 Further exploration of causal mediation will

follow the methods of Imai et al. 117, 118 We will also examine whether the effect of intervention on SFDs is mediated by provider competencies, provider/caregiver communication or caregiver self-efficacy. Missing data: Every effort to retain participants in the study will be exerted in order to avoid bias due to attrition. For those individuals who refuse continued participation, we will document reasons for study discontinuation and Rubin's multiple imputation method<sup>119</sup> with 5 repeated imputations will be employed to impute the missing endpoint for conducting the intent-to-treat analysis.

**Power Analysis.** With a recruitment of 512 participants at baseline, we anticipate a final sample of 460 participants with complete data for the primary analysis assuming no more than 10% attrition at 12 month evaluation. This estimate of attrition rate is conservative based on our prior experience. To account for the intra-cluster correlation due to cluster sampling, we estimate that an intra-provider correlation coefficient is no greater than 0.03 from our prior studies. Although the intra-practice correlation coefficient should be smaller than intra-provider correlation coefficient, we conservatively used the same value (i.e., 0.03). Under the above assumption, with 230 participants per group, we will be able to provide 80% power to detect a standardized effect size of >0.29 in change of number of SFDs. Even if actual attrition is greater than we expect (e.g., 15%), the detectable standardized effect size will only increase slightly to 0.30. Further, as we will impute missing data using informative covariates for the primary analyses, the power to detect such effects will be >80%.

Aim 3. To evaluate the process of program implementation: In order to evaluate the potential for dissemination of this primary care intervention, we will report specific summary measures recommended by the RE-AIM<sup>93</sup> framework. We will compare the provider-level proportion of visits with corrective actions taken by the eMPI providers to that of eUC providers using the same analytic approach stated in Aim 2 (Reach). We will evaluate the impact of eMPI on guideline-based corrective actions and symptoms (Effectiveness). We will qualitatively describe problem solving progress that occurs in each practice as part of process of improvement, by coding the specific barriers that arise during implementation and are collected by clinic champions, and the solutions that eMPI practices identify (Adoption). We will report consistency with which participants in the intervention arm receive the protocol through EHR data, practice observations of the process of implementation and data collected from OW contacts with participants. Additional measures of implementation of eMPI include 1) caregivers' completion of severity/control assessments at the visit; 2) provider and caregiver receipt of prompts: 3) providers' documentation of asthma discussion (Implementation). We will use provider survey responses to evaluate the extent to which each intervention component was continued or modified post-study and sustained effects on the primary outcome (Maintenance). Using EHR records of 5,000 children across all four waves of translation, we will determine if eMPI practices will (a) reach successively higher levels of guideline-based care, (b) achieve that level more guickly, and (c) sustain use of guidelines for 18 months. The analytic approach to address this will involve a statistical model with the main effect of intervention condition, time (which represents the level of Implementation), and the indicators of waves (which will allow us to evaluate sustainability), plus all the two-way and three-way interactions. We expect to see specific three-way interaction effects involving trends in rates of guideline-based care over 24 months, with an ever steeper linear increases and less pronounced downturns seen from wave to wave, in eMPI practices vs. eUC. Guidelinebased care is intended to ensure that children receive needed services in a more timely fashion. We will examine patterns of utilization by children in both groups using the EHR, including adherence to clinic visits, specialty referrals, emergency and in-patient care, and OW referrals.

# 1. Compensation

Caregivers will receive \$20 at baseline, 3, 6, and 9 months follow-up, and \$30 at 12 months follow-up. In cases where caregivers are unreachable after multiple call attempts, we will offer an additional \$10 gift card incentive in an effort to obtain accurate contact information and complete pending follow up surveys. If caregivers are still unreachable after these efforts, we will attempt to meet at the caregiver's home or in the community to complete the respective survey, obtain accurate contact information, and provide their compensation. Given the COVID-19 pandemic, as of March 2020, home visit and appointment outreach efforts have been restricted, focusing only on telephonic outreach to complete follow up surveys. In addition, each of



the 22 practices will be given a donation of \$500.00 to thank them for their participation. This participation will include providing space for research assistants to speak with families. Practice staff will also assist research staff with printing schedules and identifying families for enrollment. Providers will also be asked to complete three brief surveys: baseline, 1, and 2 year follow-ups.

There is no cost to those who participate in this study. The participants and their insurance company will be responsible for the cost of all standard of care office visits and medications. This intervention is meant only to help assure that appropriate medications are prescribed and national asthma guidelines are followed.

### 2. Safety or Risk

The study proposed should pose minimal risk to the participants, with the primary concern for loss of confidentiality. To minimize this risk, all records will be kept strictly confidential as required by the policies and procedures of the Montefiore Medical Center where data are collected, processed, or reported. Any significant concerns will be relayed promptly to the study coordinator, the principal investigator, the NHLBI, and the Institutional Review Board. During follow-up, all children with persistent symptoms or poor control will be referred to their primary care provider for care. The primary care provider or the family can discontinue the child's participation at any time during the study.

#### 3. Data Storage and Confidentiality

Recruitment, Informed Consent, and Confidentiality: Human subjects' rights will be protected as explained in the consent form used for the study. The Institutional Review Board (IRB) will review all protocol and informed consent documents and research will be carried out only after proper approval from the IRB. Written consent will be obtained prior to the initiation of any research evaluations from the subset of 512 participants. Informed consent will be obtained from all potential subjects by a researcher trained and certified in human subjects protection. The informed consent process will detail the potential benefits of participating in the research as well as the potential risks of the intervention. Assent also will be obtained from children in the program who are 7 years of age and older. Subjects will be informed that they may choose not to answer any of the questions on the surveys and that they may withdraw from the study at any time without negative consequences. Strict confidentiality will be maintained throughout the study. The data will be stored in password protected computers and locked file cabinets in a study office, and only the researchers or their associates will have access to these data.

We will obtain a waiver of consent to be able to review de-identified EHR data by practice to identify the proportion of visits with > 1 guideline-based corrective actions (clinic-level variable). These data will be obtained on a clinic-level without identifying specific patients.

To obtain a waiver of consent, the following criteria will be met (45 CFR 46.116(d):

- (1) The research involves no more than minimal risk to the subjects:
- (2) The waiver or alteration will not adversely affect the rights and welfare of the subjects:
- (3) The research could not practicably be carried out without the waiver or alteration; and
- (4) Whenever appropriate, the subjects will be provided with additional pertinent information after participation.

#### Protection against Risk:

During recruitment, parents will be offered private areas in the waiting room to conduct informed consent and baseline assessments. For confidentiality protection, the identity and personal information of each subject will be used only for purposes of this study and will only be accessed by appropriate study personnel. For specific analyses, files consisting of pertinent data from the individual records will be formed from the base data file. All data will be held confidentially and stored in locked files, accessible to authorized staff and investigators only.

Any parent indicating high risk for depression during a follow-up interview will be referred to their primary care provider or mental health provider present in each clinic, and will be sent a summary of community resources available for care. Additionally, parents will be informed of emergency resources at the time of the telephone interview, including lifeline, social work supports, and 911. This mechanism is being used in our current

school-based study, is approved by our institutional review board, and has been well received by parents. Additional Measures to Protect the Data:

We will take additional measures to minimize the risk of breaching the confidentiality of data. These include but are not limited to the following:

- Electronic firewalls
- Audit trails
- Disaster prevention and recovery plans
- Systems certification
- All research personnel take yearly HIPAA training

Identity of participants will not be revealed in the presentation or publication of any results from the project. All personnel working on the project will be regularly educated about the importance of strictly respecting participants' rights to confidentiality.

# **Data and Safety Monitoring Plan**

## **Data Quality Monitoring**

Baseline data forms will be completed electronically by research staff on Tablet PCs in the waiting room. All survey data collected on the Tablet PCs are entered using data entry forms created by Adobe Creative Suite 3 software, which allows for integration with secure data entry forms to an off-site server. Asthma severity and control assessment and data necessary for generation of the prompts will be entered into each patient's EPIC Electronic Health Record (EHR). For the safety of private subject information, no data will be stored on the Tablet PCs. For the 4 follow-up telephone interviews, data will be collected using RedCap database. Pre-intervention training of study staff will be conducted to increase knowledge about asthma, asthma medications, and other important information in order to reduce the number of "real-time" data collection errors. Through this training, staff will note any inconsistencies in parent reported data and will discuss them with the parent at the time of the interview.

A separate team of researchers will perform all follow-up interviews and follow-up data management. This group will work independently from the "enrollment team" and thus will be able to perform blinded assessments of outcomes. Randomization information will not be included with any follow-up materials in order to assure blinding of outcome assessment.

Once data have been collected, simple range checks as well as cross-form validation checks will be performed to ensure the accuracy and completeness of the data. A list of all data checks performed will be maintained and any errors detected by this method will be noted. In addition, data forms, valid informed consent documents for each enrolled patient, and supporting source documentation materials will be reviewed by the data analysts for accuracy. Required regulatory documents (IRB approval, updates to the protocol, data monitoring documents) will be maintained by the study coordinator. All events during the course of the trial including study enrollments, adverse events and study terminations will be reported to the study coordinator (see safety section below).

# Safety Monitoring Plan

Potential risks related to participation in this study are minimal since surveys are administered and information is relayed to caregivers and providers during the time that children will be receiving care at their primary care office. No medications or investigational treatments are given as part of this study. Any significant adverse events will be flagged by the follow-up team and relayed promptly to the study coordinator, the principal investigator, the child's primary care provider, and the Institutional Review Board within 24 hours. We plan to hold monthly research review meetings with the study team to provide monitoring to ensure subject safety as well as treatment integrity. Any child experiencing an exacerbation or persistent symptoms at the time of an assessment will be referred to their primary care provider. All records will be kept strictly confidential as required by the policies and procedures of the Albert Einstein College of Medicine /Montefiore Medical Center

where data are collected, processed, or reported. The family can discontinue their participation at any time during the study.

### 4. Potential Benefits

There are potential benefits of this intervention. Children obtaining care from the eMPI practices may have improved care due to the use of prompts and telephone-based care coordination, education and support provided by the Outreach Worker to help promote discussion of the child's asthma, provide recommendations for asthma care and promote full adoption of asthma guidelines. In addition, both groups may benefit by having the asthma guidelines reinforced with all practices, and providing resources for physicians. All families will receive multiple phone calls in order to assess the child's symptoms. It is possible that an increased awareness of symptoms and enhanced communication with the primary care provider will occur, and will result in reduced morbidity for these children.

## **Bibliography & References Cited**

- 1. Bloom B, Jones LI, Freeman G. Summary health statistics for U.S. children: National Health Interview Survey, 2012. National Center for Health Statistics. Vital Health Stat 2013;10:1-81.
- 2. Flores G, Snowden-Bridon C, Torres S, Perez R, Walter T, Brotanek J, Lin H, Tomany-Korman S. Urban minority children with asthma: substantial morbidity, compromised quality and access to specialists, and the importance of poverty and specialty care. *J Asthma*. 2009;46(4):392-398.
- Szefler SJ, Mitchell H, Sorkness CA, Gergen PJ, O'Connor GT, Morgan WJ, Kattan M, Pongracic JA, Teach SJ, Bloomberg GR, Eggleston PA, Gruchalla RS, Kercsmar CM, Liu AH, Wildfire JJ, Curry MD, Busse WW. Management of asthma based on exhaled nitric oxide in addition to guideline-based treatment for inner-city adolescents and young adults: a randomised controlled trial. *Lancet*. 2008;372(9643):1065-1072.
- 4. Wisnivesky JP, Lorenzo J, Lyn-Cook R, Newman T, Aponte A, Kiefer E, Halm EA. Barriers to adherence to asthma management guidelines among inner-city primary care providers. *Ann Allergy Asthma Immunol*. 2008;101(3):264-270.
- 5. Okelo SO, Butz AM, Sharma R, Diette GB, Pitts SI, King TM, Linn ST, Reuben M, Chelladurai Y, Robinson KA. Interventions to modify health care provider adherence to asthma guidelines: a systematic review. *Pediatrics*. 2013;132(3):517-534.
- 6. Cabana MD, Rand CS, Powe NR, Wu AW, Wilson MH, Abboud PA, Rubin HR. Why don't physicians follow clinical practice guidelines? A framework for improvement. *JAMA*. 1999;282(15):1458-1465.
- 7. Cabana MD, Ebel BE, Cooper-Patrick L, Powe NR, Rubin HR, Rand CS. Barriers pediatricians face when using asthma practice guidelines. *Arch Pediatr Adolesc Med*. 2000;154(7):685-693.
- 8. Frey SM, Fagnano M, Halterman JS. Caregiver education to promote appropriate use of preventive asthma medications: what is happening in primary care? *J Asthma*. 2015:1-7.
- Okelo SO, Butz AM, Sharma R, Diette GB, Pitts SI, King TM, Linn ST, Reuben M, Chelladurai Y, Robinson KA. Interventions to Modify Health Care Provider Adherence to Asthma Guidelines. AHRQ Comparative Effectiveness Review. May 2013. AHRQ Pub. No. 13-EHC022-1-EF. www.effectivehealthcare.ahrq.gov/reports/final.cfm Accessed October 5, 2015.
- 10. Reznik M, Jaramillo Y, Wylie-Rosett J. Demonstrating and assessing metered-dose inhaler-spacer technique: pediatric care providers' self-reported practices and perceived barriers. *Clin Pediatr (Phila)*. 2014;53(3):270-276.
- 11. Okelo SO, Siberry GK, Solomon BS, Bilderback AL, Yamazaki M, Hetzler T, Ferrell CL, Dhepyasuwan N, Serwint JR, Investigators C. Asthma treatment decisions by pediatric residents do not consistently conform to guidelines or improve with level of training. *Acad Pediatr*. 2014;14(3):287-293.
- 12. Shiffman RN, Freudigman M, Brandt CA, Liaw Y, Navedo DD. A guideline implementation system using handheld computers for office management of asthma: effects on adherence and patient outcomes. *Pediatrics*. 2000;105(4 Pt 1):767-773.
- 13. Cloutier MM, Wakefield DB, Carlisle PS, Bailit HL, Hall CB. The effect of Easy Breathing on asthma management and knowledge. *Arch Pediatr Adolesc Med.* 2002;156(10):1045-1051.
- 14. Eccles M, McColl E, Steen N, Rousseau N, Grimshaw J, Parkin D, Purves I. Effect of computerised evidence based guidelines on management of asthma and angina in adults in primary care: cluster randomised controlled trial. *BMJ*. 2002;325(7370):941.
- 15. Cloutier MM, Hall CB, Wakefield DB, Bailit H. Use of asthma guidelines by primary care providers to reduce hospitalizations and emergency department visits in poor, minority, urban children. *J Pediatr*. 2005;146(5):591-597.
- 16. Lesho EP, Myers CP, Ott M, Winslow C, Brown JE. Do clinical practice guidelines improve processes or outcomes in primary care? *Mil Med*. 2005;170(3):243-246.
- 17. Mitchell EA, Didsbury PB, Kruithof N, Robinson E, Milmine M, Barry M, Newman J. A randomized controlled trial of an asthma clinical pathway for children in general practice. *Acta Paediatr*. 2005;94(2):226-233.

- 18. Halterman JS, Fisher S, Conn KM, Fagnano M, Lynch K, Marky A, Szilagyi PG. Improved preventive care for asthma: a randomized trial of clinician prompting in pediatric offices. *Arch Pediatr Adolesc Med*. 2006;160(10):1018-1025.
- 19. Martens JD, van der Weijden T, Severens JL, de Clercq PA, de Bruijn DP, Kester AD, Winkens RA. The effect of computer reminders on GPs' prescribing behaviour: a cluster-randomised trial. *Int J Med Inform*. 2007;76 Suppl 3:S403-416.
- 20. Bell LM, Grundmeier R, Localio R, Zorc J, Fiks AG, Zhang X, Stephens TB, Swietlik M, Guevara JP. Electronic health record-based decision support to improve asthma care: a cluster-randomized trial. *Pediatrics*. 2010;125(4):e770-777.
- 21. Cho SH, Jeong JW, Park HW, Pyun BY, Chang SI, Moon HB, Kim YY, Choi BW. Effectiveness of a computer-assisted asthma management program on physician adherence to guidelines. *J Asthma*. 2010;47(6):680-686.
- Davis AM, Cannon M, Ables AZ, Bendyk H. Using the electronic medical record to improve asthma severity documentation and treatment among family medicine residents. Fam Med. 2010;42(5):334-337.
- de Vries TW, van den Berg PB, Duiverman EJ, de Jong-van den Berg LT. Effect of a minimal pharmacy intervention on improvement of adherence to asthma guidelines. *Arch Dis Child*. 2010;95(4):302-304.
- 24. Ragazzi H, Keller A, Ehrensberger R, Irani AM. Evaluation of a practice-based intervention to improve the management of pediatric asthma. *J Urban Health*. 2011;88 Suppl 1:38-48.
- 25. Gupta RS, Weiss KB. The 2007 National Asthma Education and Prevention Program asthma guidelines: accelerating their implementation and facilitating their impact on children with asthma. *Pediatrics*. 2009;123 Suppl 3:S193-198.
- 26. Shapiro A, Gracy D, Quinones W, Applebaum J, Sarmiento A. Putting guidelines into practice: improving documentation of pediatric asthma management using a decision-making tool. *Arch Pediatr Adolesc Med.* 2011;165(5):412-418.
- 27. Wagner EH, Austin BT, Davis C, Hindmarsh M, Schaefer J, Bonomi A. Improving chronic illness care: translating evidence into action. *Health Aff (Millwood)*. 2001;20(6):64-78.
- 28. Halterman JS, Fagnano M, Tremblay PJ, Fisher SG, Wang H, Rand C, Szilagyi P, Butz A. Prompting asthma intervention in Rochester-uniting parents and providers (PAIR-UP): a randomized trial. *JAMA Pediatr*. 2014;168(10):e141983.
- 29. Garg R, Karpati A, Leighton J, Perrin M, Shah M. Asthma Facts, Second Edition. New York City Department of Health and Mental Hygiene. May 2003. Available at: <a href="http://www.nyc.gov/html/doh/downloads/pdf/asthma/facts.pdf">http://www.nyc.gov/html/doh/downloads/pdf/asthma/facts.pdf</a>. Accessed June 11, 2015.
- 30. Smith LA, Hatcher-Ross JL, Wertheimer R, Kahn RS. Rethinking race/ethnicity, income, and childhood asthma: racial/ethnic disparities concentrated among the very poor. *Public Health Rep.* 2005;120:109-116.
- 31. Claudio L, Stingone JA, Godbold J. Prevalence of childhood asthma in urban communities: the impact of ethnicity and income. *Ann Epidemiol*. 2006;16(5):332-340.
- 32. Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007 *Pediatrics*. 2009;123:S131-S145.
- 33. Bloom B, Cohen RA, Freeman G. Summary health statistics for US children: National Health Interview Survey, 2007 *Vital Health Stat.* 2009;10(239):1-88.
- 34. Cabana MD, Lara M, Shannon J. Racial and ethnic disparities in the quality of asthma care. *Chest.* 2007;132(5 Suppl):810S-817S.
- 35. Webber MP, Carpiniello KE, Oruwariye T, Lo Y, Burton WB, Appel DK. Burden of asthma in inner-city elementary schoolchildren: do school-based health centers make a difference? *Arch Pediatr Adolesc Med.* 2003;157(2):125-129.
- 36. Reznik M, Bauman LJ, Okelo SO, Halterman JS. Asthma identification and medication administration forms in New York City schools. *Ann Allergy Asthma Immunol*. 2015;114(1):67-68 e61.
- 37. Wu AC, Smith L, Bokhour B, Hohman KH, Lieu TA. Racial/Ethnic variation in parent perceptions of asthma. *Ambul Pediatr*. 2008;8(2):89-97.

- 38. Halterman JS, Auinger P, Conn KM, Lynch K, Yoos HL, Szilagyi PG. Inadequate therapy and poor symptom control among children with asthma: findings from a multistate sample. *Ambul Pediatr*. 2007;7(2):153-159.
- 39. Akinbami LJ, Moorman JE, Simon AE, Schoendorf KC. Trends in racial disparities for asthma outcomes among children 0 to 17 years, 2001-2010. *J Allergy Clin Immunol*. 2014;134(3):547-553 e545.
- 40. Capo-Ramos DE, Duran C, Simon AE, Akinbami LJ, Schoendorf KC. Preventive asthma medication discontinuation among children enrolled in fee-for-service Medicaid. *J Asthma*. 2014;51(6):618-626.
- 41. National Heart Lung and Blood Institute. National Asthma Education and Prevention Program. Expert panel report 3: guidelines for the diagnosis and management of asthma. NIH Publication Number 08-5846. Bethesda, MD: 2007. http://www.nhlbi.nih.gov/guidelines/asthma/ Accessed October 5, 2015.
- 42. Cabana MD, Bruckman D, Meister K, Bradley JF, Clark N. Documentation of asthma severity in pediatric outpatient clinics. *Clin Pediatr (Phila)*. 2003;42(2):121-125.
- 43. Biksey T, Zickmund S, Wu F. Disparities in risk communication: a pilot study of asthmatic children, their parents, and home environments. *J Natl Med Assoc.* 2011;103(5):388-391.
- Bousquet J, Khaltaev N, Cruz AA, Denburg J, Fokkens WJ, Togias A, Zuberbier T, Baena-Cagnani CE, 44. Canonica GW, van Weel C, Agache I, Ait-Khaled N, Bachert C, Blaiss MS, Bonini S, Boulet LP, Bousquet PJ, Camargos P, Carlsen KH, Chen Y, Custovic A, Dahl R, Demoly P, Douagui H, Durham SR. van Wijk RG. Kalavci O. Kaliner MA. Kim YY. Kowalski ML. Kuna P. Le LT. Lemiere C. Li J. Lockev RF, Mavale-Manuel S, Meltzer EO, Mohammad Y, Mullol J, Naclerio R, O'Hehir RE, Ohta K, Ouedraogo S, Palkonen S, Papadopoulos N, Passalacqua G, Pawankar R, Popov TA, Rabe KF, Rosado-Pinto J, Scadding GK, Simons FE, Toskala E, Valovirta E, van Cauwenberge P, Wang DY, Wickman M, Yawn BP, Yorgancioglu A, Yusuf OM, Zar H, Annesi-Maesano I, Bateman ED, Ben Kheder A, Boakye DA, Bouchard J, Burney P, Busse WW, Chan-Yeung M, Chavannes NH, Chuchalin A, Dolen WK, Emuzyte R, Grouse L, Humbert M, Jackson C, Johnston SL, Keith PK, Kemp JP, Klossek JM, Larenas-Linnemann D, Lipworth B, Malo JL, Marshall GD, Naspitz C, Nekam K, Niggemann B, Nizankowska-Mogilnicka E, Okamoto Y, Orru MP, Potter P, Price D, Stoloff SW, Vandenplas O, Viegi G, Williams D, World Health O, Galen, AllerGen. Allergic Rhinitis and its Impact on Asthma (ARIA) 2008 update (in collaboration with the World Health Organization, GA(2)LEN and AllerGen). Allergy. 2008;63 Suppl 86:8-160.
- 45. Diaz J, Farzan S. Clinical implications of the obese-asthma phenotypes. *Immunol Allergy Clin North Am*. 2014;34(4):739-751.
- 46. Scadding G, Walker S. Poor asthma control?--then look up the nose. The importance of co-morbid rhinitis in patients with asthma. *Prim Care Respir J.* 2012;21(2):222-228.
- 47. Lee MG, Cross KJ, Yang WY, Sutton BS, Jiroutek MR. Frequency of asthma education in primary care in the years 2007-2010. *J Asthma*. 2015:1-7.
- 48. McMullen A, Yoos HL, Anson E, Kitzmann H, Halterman JS, Arcoleo KS. Asthma care of children in clinical practice: do parents report receiving appropriate education? *Pediatr Nurs*. 2007;33(1):37-44.
- 49. Reznik M, Silver EJ, Cao Y. Evaluation of MDI-spacer utilization and technique in caregivers of urban minority children with persistent asthma. *J Asthma*. 2014;51(2):149-154.
- 50. Conn KM, Halterman JS, Lynch K, Cabana MD. The impact of parents' medication beliefs on asthma management. *Pediatrics*. 2007;120(3):e521-526.
- 51. Mitchell SJ, Bilderback AL, Okelo SO. Racial Disparities in Asthma Morbidity Among Pediatric Patients Seeking Asthma Specialist Care. *Acad Pediatr.* 2015.
- 52. James CV, Rosenbaum S. Paying for quality care: implications for racial and ethnic health disparities in pediatric asthma. *Pediatrics*. 2009;123 Suppl 3:S205-210.
- 53. Tsuyuki RT, Sin DD, Sharpe HM, Cowie RL, Nilsson C, Man SF. Management of asthma among community-based primary care physicians. *J Asthma*. 2005;42(3):163-167.
- 54. Powell BJ, Waltz TJ, Chinman MJ, Damschroder LJ, Smith JL, Matthieu MM, Proctor EK, Kirchner JE. A refined compilation of implementation strategies: results from the Expert Recommendations for Implementing Change (ERIC) project. *Implement Sci.* 2015;10:21.
- 55. Butz AM, Walker J, Land CL, Vibbert C, Winkelstein M. Improving asthma communication in high-risk children. *J Asthma*. 2007;44(9):739-745.



- 56. Kattan M, Crain EF, Steinbach S, Visness CM, Walter M, Stout JW, Evans R, 3rd, Smartt E, Gruchalla RS, Morgan WJ, O'Connor GT, Mitchell HE. A randomized clinical trial of clinician feedback to improve quality of care for inner-city children with asthma. *Pediatrics*. 2006;117(6):e1095-1103.
- 57. Vernacchio L, Francis ME, Epstein DM, Santangelo J, Trudell EK, Reynolds ME, Risko W. Effectiveness of an asthma quality improvement program designed for maintenance of certification. *Pediatrics*. 2014;134(1):e242-248.
- 58. Richman MJ, Poltawsky JS. Partnership for excellence in asthma care: evidence-based disease management. *Stud Health Technol Inform*. 2000;76:107-121.
- 59. Baker R, Fraser RC, Stone M, Lambert P, Stevenson K, Shiels C. Randomised controlled trial of the impact of guidelines, prioritized review criteria and feedback on implementation of recommendations for angina and asthma. *Br J Gen Pract*. 2003;53(489):284-291.
- 60. Coleman CI, Reddy P, Laster-Bradley NM, Dorval S, Munagala B, White CM. Effect of practitioner education on adherence to asthma treatment guidelines. *Ann Pharmacother*. 2003;37(7-8):956-961.
- 61. Schneider A, Wensing M, Biessecker K, Quinzler R, Kaufmann-Kolle P, Szecsenyi J. Impact of quality circles for improvement of asthma care: results of a randomized controlled trial. *J Eval Clin Pract*. 2008;14(2):185-190.
- 62. Daniels EC, Bacon J, Denisio S, Fry YW, Murray V, Quarshie A, Rust G. Translation squared: improving asthma care for high-disparity populations through a safety net practice-based research network. *J Asthma*. 2005;42(6):499-505.
- 63. Frankowski BL, Keating K, Rexroad A, Delaney T, McEwing SM, Wasko N, Lynn S, Shaw J. Community collaboration: concurrent physician and school nurse education and cooperation increases the use of asthma action plans. *J Sch Health*. 2006;76(6):303-306.
- 64. Yawn BP, Bertram S, Wollan P. Introduction of Asthma APGAR tools improve asthma management in primary care practices. *J Asthma Allergy*. 2008;1:1-10.
- 65. Bender BG, Dickinson P, Rankin A, Wamboldt FS, Zittleman L, Westfall JM. The Colorado Asthma Toolkit Program: a practice coaching intervention from the High Plains Research Network. *J Am Board Fam Med*. 2011;24(3):240-248.
- 66. Lob SH, Boer JH, Porter PG, Nunez D, Fox P. Promoting best-care practices in childhood asthma: quality improvement in community health centers. *Pediatrics*. 2011;128(1):20-28.
- 67. Evans D, Sheares BJ, Vazquez TL. Educating health professionals to improve quality of care for asthma. *Paediatr Respir Rev.* 2004;5(4):304-310.
- 68. Lozano P, Finkelstein JA, Carey VJ, Wagner EH, Inui TS, Fuhlbrigge AL, Soumerai SB, Sullivan SD, Weiss ST, Weiss KB. A multisite randomized trial of the effects of physician education and organizational change in chronic-asthma care: health outcomes of the Pediatric Asthma Care Patient Outcomes Research Team II Study. *Arch Pediatr Adolesc Med.* 2004;158(9):875-883.
- 69. Glasgow RE, Nutting PA, King DK, Nelson CC, Cutter G, Gaglio B, Rahm AK, Whitesides H, Amthauer H. A practical randomized trial to improve diabetes care. *J Gen Intern Med*. 2004;19(12):1167-1174.
- 70. Tunis SR, Stryer DB, Clancy CM. Practical clinical trials: increasing the value of clinical research for decision making in clinical and health policy. *Jama*. 2003;290(12):1624-1632.
- 71. Smedley BD, Stith AY, Nelson AR, eds. Unequal Treatment: Confronting Racial and Ethnic Disparities in Health Care. Washington, DC: National Academies Press, 2002.
- 72. Mason T, Wilkinson GW, Nannini A, Martin CM, Fox DJ, Hirsch G. Winning policy change to promote community health workers: lessons from massachusetts in the health reform era. *Am J Public Health*. 2011;101(12):2211-2216.
- 73. Margellos-Anast H, Gutierrez MA, Whitman S. Improving asthma management among African-American children via a community health worker model: findings from a Chicago-based pilot intervention. *J Asthma*. 2012;49(4):380-389.
- 74. Campbell JD, Brooks M, Hosokawa P, Robinson J, Song L, Krieger J. Community Health Worker Home Visits for Medicaid-Enrolled Children With Asthma: Effects on Asthma Outcomes and Costs. *Am J Public Health*. 2015;105(11):2366-2372.

- 75. Reznik M, Silver EJ, Jaramillo Y. A Randomized Trial of a Community Health Worker (CHW) Led Asthma Intervention: Preliminary Findings. 2014 Pediatric Academic Societies and Asian Society for Pediatric Research Joint Meeting, Vancouver, BC, Canada May 3-6, 2014.
- 76. Peretz PJ, Matiz LA, Findley S, Lizardo M, Evans D, McCord M. Community health workers as drivers of a successful community-based disease management initiative. *Am J Public Health*. 2012;102(8):1443-1446.
- 77. Fisher-Owens SA, Boddupalli G, Thyne SM. Telephone case management for asthma: an acceptable and effective intervention within a diverse pediatric population. *J Asthma*. 2011;48(2):156-161.
- 78. Garbutt JM, Sylvia S, Rook S, Schmandt M, Ruby-Ziegler C, Luby J, Strunk RC. Peer training to improve parenting and childhood asthma management skills: a pilot study. *Ann Allergy Asthma Immunol*. 2015;114(2):148-149.
- 79. Garbutt JM, Yan Y, Highstein G, Strunk RC. A cluster-randomized trial shows telephone peer coaching for parents reduces children's asthma morbidity. *J Allergy Clin Immunol*. 2015;135(5):1163-1170 e1161-1162.
- 80. Patient-Centered Medical Home Recognition.

  <a href="http://www.ncqa.org/Programs/Recognition/Practices/PatientCenteredMedicalHomePCMH.aspx">http://www.ncqa.org/Programs/Recognition/Practices/PatientCenteredMedicalHomePCMH.aspx</a>

  Accessed October 10, 2015.
- 81. Thorpe KE, Zwarenstein M, Oxman AD, Treweek S, Furberg CD, Altman DG, Tunis S, Bergel E, Harvey I, Magid DJ, Chalkidou K. A pragmatic-explanatory continuum indicator summary (PRECIS): a tool to help trial designers. *CMAJ*. 2009;180(10):E47-57.
- 82. Rapkin BD, Weiss ES, Lounsbury DW, Thompson HS, Goodman RM, Schechter CB, Merzel C, Shelton RC, Blank AE, Erb-Downward J, Williams A, Valera P, Padgett DK. Using the interactive systems framework to support a quality improvement approach to dissemination of evidence-based strategies to promote early detection of breast cancer: planning a comprehensive dynamic trial. *Am J Community Psychol.* 2012;50(3-4):497-517.
- 83. Rapkin B.D., Trickett E.J. Comprehensive Dynamic Trial Designs for Behavioral Prevention Research with Communities: Overcoming Inadequacies of the Randomized Controlled Trial Paradigm. In Community Interventions and AIDS. Eds. Trickett E.J. and Pequegnat W. Oxford University Press. 2005:249-277.
- 84. Reznik M, Bauman LJ. Barriers to Physical Activity in Schoolchildren with Asthma: A Parent Perspective *Clinical and Translational Science* 2012;5(2):168.
- 85. Brown JV, Bakeman R, Celano MP, Demi AS, Kobrynski L, Wilson SR. Home-based asthma education of young low-income children and their families. *J Pediatr Psychol*. 2002;27(8):677-688.
- 86. Reznik M, Wylie-Rosett J, Kim M, Ozuah PO. A Classroom-Based Physical Activity Intervention for Urban Kindergarten and First-Grade Students: A Feasibility Study. *Childhood Obesity*. 2015;11(3):314-324.
- 87. Halterman JS, Riekert K, Bayer A, Fagnano M, Tremblay P, Blaakman S, Borrelli B. A pilot study to enhance preventive asthma care among urban adolescents with asthma. *J Asthma*. 2011;48(5):523-530.
- 88. Halterman JS, Szilagyi PG, Fisher SG, Fagnano M, Tremblay P, Conn KM, Wang H, Borrelli B. Randomized controlled trial to improve care for urban children with asthma: results of the School-Based Asthma Therapy trial. *Arch Pediatr Adolesc Med.* 2011;165(3):262-268.
- 89. Rinke ML, Chen AR, Bundy DG, Colantuoni E, Fratino L, Drucis KM, Panton SY, Kokoszka M, Budd AP, Milstone AM, Miller MR. Implementation of a central line maintenance care bundle in hospitalized pediatric oncology patients. *Pediatrics*. 2012;130(4):e996-e1004.
- 90. Rinke ML, Dietrich E, Kodeck T, Westcoat K. Operation care: a pilot case management intervention for frequent emergency medical system users. *Am J Emerg Med*. 2012;30(2):352-357.
- 91. Basu Roy U, Michel T, Carpenter A, Lounsbury DW, Sabino E, Stevenson AJ, Combs S, Jacobs J, Padgett D, Rapkin BD. Community-led cancer action councils in Queens, New York: process evaluation of an innovative partnership with the Queens library system. *Prev Chronic Dis.* 2014;11:130176.



- 92. Blaakman S, Tremblay PJ, Halterman JS, Fagnano M, Borrelli B. Implementation of a communitybased secondhand smoke reduction intervention for caregivers of urban children with asthma: process evaluation, successes and challenges. Health Educ Res. 2013;28(1):141-152.
- 93. Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. *Am J Public Health*. 1999;89(9):1322-1327.
- 94. Wagner EH. Chronic disease management: what will it take to improve care for chronic illness? Eff Clin Pract. 1998;1(1):2-4.
- Ockene JK. Zapka JG. Provider education to promote implementation of clinical practice guidelines. 95. Chest. 2000;118(2 Suppl):33s-39s.
- 96. RE-AIM Planning Tool. http://www.re-aim.hnfe.vt.edu/forms/re-aim planning tool and adaptation.pdf Accessed on October 19, 2015.
- 97. Soumerai SB, Avorn J. Principles of educational outreach ('academic detailing') to improve clinical decision making. Jama. 1990;263(4):549-556.
- 98. Halterman JS, McConnochie KM, Conn KM, Yoos HL, Callahan PM, Neely TL, Szilagyi PG. A randomized trial of primary care provider prompting to enhance preventive asthma therapy. Arch Pediatr Adolesc Med. 2005;159(5):422-427.
- Cabana MD, Slish KK, Evans D, Mellins RB, Brown RW, Lin X, Kaciroti N, Clark NM. Impact of 99. Physician Asthma Care Education on patient outcomes. Health Educ Behav. 2014;41(5):509-517.
- 100. Allen FC, Vargas PA, Kolodner K, Eggleston P, Butz A, Huss K, Malveaux F, Rand CS. Assessing pediatric clinical asthma practices and perceptions: a new instrument. J Asthma. 2000;37(1):31-42.
- 101. Cabana MD, Slish KK, Evans D, Mellins RB, Brown RW, Lin X, Kaciroti N, Clark NM, Impact of physician asthma care education on patient outcomes. *Pediatrics*. 2006;117(6):2149-2157.
- 102. Clark NM, Gong M, Schork MA, Maiman LA, Evans D, Hurwitz ME, Roloff D, Mellins RB. A scale for Assessing Health Care Providers' Teaching and Communication Behavior regarding asthma. Health Educ Behav. 1997;24(2):245-256.
- Reddel HK, Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, Casale TB, Chanez P, 103. Enright PL, Gibson PG, de Jongste JC, Kerstjens HA, Lazarus SC, Levy ML, O'Byrne PM, Partridge MR, Pavord ID, Sears MR, Sterk PJ, Stoloff SW, Sullivan SD, Szefler SJ, Thomas MD, Wenzel SE, American Thoracic Society/European Respiratory Society Task Force on Asthma C, Exacerbations. An official American Thoracic Society/European Respiratory Society statement: asthma control and exacerbations: standardizing endpoints for clinical asthma trials and clinical practice. Am J Respir Crit Care Med. 2009:180(1):59-99.
- 104. Busse WW, Morgan WJ, Taggart V, Togias A. Asthma outcomes workshop: overview. J Allergy Clin Immunol. 2012;129(3 Suppl):S1-8.
- 105. Schatz M, Zeiger RS, Drane A, Harden K, Cibildak A, Oosterman JE, Kosinski M. Reliability and predictive validity of the Asthma Control Test administered by telephone calls using speech recognition technology. J Allergy Clin Immunol. 2007;119(2):336-343.
- 106. Juniper EF, Guyatt GH, Feeny DH, Ferrie PJ, Griffith LE, Townsend M. Measuring quality of life in the parents of children with asthma. Qual Life Res. 1996;5(1):27-34.
- 107. Asmussen L, Olson LM, Grant EN, Fagan J, Weiss KB. Reliability and validity of the Children's Health Survey for Asthma. *Pediatrics*. 1999:104(6):e71.
- 108. Horne R WJ HM. The beliefs about medicines questionnaire: The development and evaluation of a new method for assessing the cognitive representation of medication. Psych Health. 1999.
- 109. Pak L, Allen PJ. The impact of maternal depression on children with asthma. *Pediatr Nurs*. 2012;38(1):11-19, 30.
- 110. Otsuki M, Eakin MN, Arceneaux LL, Rand CS, Butz AM, Riekert KA. Prospective relationship between maternal depressive symptoms and asthma morbidity among inner-city African American children. J Pediatr Psychol. 2010;35(7):758-767.
- 111. Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001;16(9):606-613.
- 112. Clark NM, Gong M, Schork MA, Evans D, Roloff D, Hurwitz M, Maiman L, Mellins RB. Impact of education for physicians on patient outcomes. *Pediatrics*. 1998;101(5):831-836.



- 113. Maly RC, Leake B, Silliman RA. Breast cancer treatment in older women: impact of the patient-physician interaction. *J Am Geriatr Soc.* 2004;52(7):1138-1145.
- 114. Maly RC, Leake B, Silliman RA. Health care disparities in older patients with breast carcinoma: informational support from physicians. *Cancer*. 2003;97(6):1517-1527.
- 115. Maly RC, Frank JC, Marshall GN, DiMatteo MR, Reuben DB. Perceived efficacy in patient-physician interactions (PEPPI): validation of an instrument in older persons. *J Am Geriatr Soc.* 1998;46(7):889-894.
- 116. MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. *Psychol Methods*. 2002;7(1):83-104.
- 117. Imai K, Keele L, Tingley D. A general approach to causal mediation analysis. *Psychol Methods*. 2010;15(4):309-334.
- 118. Imai K, Keele L, Tingley D, Yamamoto T (2010). Causal Mediation Analysis Using R." In HD Vinod (ed.), Advances in Social Science Research Using R, Lecture Notes in Statistics, pp. 129{154. Springer-Verlag, New York.
- 119. Rubin, D.B. (1976) Inference and missing data. Biometrika, 63, 581-592.
- 120. Finkelstein JA, Lozano P, Streiff KA, Arduino KE, Sisk CA, Wagner EH, Weiss KB, Inui TS. Clinical effectiveness research in managed-care systems: lessons from the Pediatric Asthma Care PORT. Patient Outcomes Research Team. *Health Serv Res.* 2002;37(3):775-789.
- 121. Fuhlbrigge AL, Kitch BT, Paltiel AD, Kuntz KM, Neumann PJ, Dockery DW, Weiss ST. FEV(1) is associated with risk of asthma attacks in a pediatric population. *J Allergy Clin Immunol*. 2001;107(1):61-67.
- 122. Jenkins HA, Cherniack R, Szefler SJ, Covar R, Gelfand EW, Spahn JD. A comparison of the clinical characteristics of children and adults with severe asthma. *Chest*. 2003;124(4):1318-1324.
- 123. Sharek PJ, Mayer ML, Loewy L, Robinson TN, Shames RS, Umetsu DT, Bergman DA. Agreement among measures of asthma status: a prospective study of low-income children with moderate to severe asthma. *Pediatrics*. 2002;110(4):797-804.
- 124. Bacharier LB MD, Lemanske RF, Schend V, Sorkness C, Strunk RC. Classifying asthma severity in children: is measuring lung function helpful? . *J Allergy Clin Immunol*. 2002.
- 125. Spahn JD, Cherniack R, Paull K, Gelfand EW. Is forced expiratory volume in one second the best measure of severity in childhood asthma? *Am J Respir Crit Care Med*. 2004;169(7):784-786.